CLINICAL TRIAL: NCT00353938
Title: Phase II Pilot Randomized Double-Blind Placebo-Controlled Study of 3,4-methylenedioxymethamphetamine (MDMA)Assisted Psychotherapy in Posttraumatic Stress Disorder (PTSD)- Switzerland
Brief Title: Study of 3,4-Methylenedioxymethamphetamine-assisted Psychotherapy in People With Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Collaborators: Swiss Medical Society for Psycholytic Therapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-2
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD, MDMA, psychotherapy, Switzerland
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Dose MDMA-assisted therapy (125 mg) (Experimental): Three 8-hour sessions of MDMA-assisted therapy with 125 mg of MDMA, followed by a supplemental dose of 62.5 mg MDMA
  Interventions: Drug: 3,4-methylenedioxymethamphetamine (125 mg); Behavioral: Therapy
- Active Placebo MDMA-assisted therapy (25 mg) (Active Comparator): Three 8-hour sessions of MDMA-assisted therapy with 25 mg of MDMA, followed by a supplemental dose of 12.5 mg MDMA
  Interventions: Drug: 3,4-methyelendioxymethamphetamine (25 mg); Behavioral: Therapy

INTERVENTIONS:
Drug: 3,4-methylenedioxymethamphetamine (125 mg) — Participants will receive an initial dose of 125 mg MDMA orally and, if investigator and participant deem appropriate, 2.5 hours later they will receive 62.5 mg MDMA orally.
  Other Names: MDMA
  Arms: Full Dose MDMA-assisted therapy (125 mg)
Drug: 3,4-methyelendioxymethamphetamine (25 mg) — Participants will receive a 25 mg MDMA orally, and if investigator and participant agree, 2.5 hours later they will receive 12.5 mg MDMA orally.
  Other Names: MDMA
  Arms: Active Placebo MDMA-assisted therapy (25 mg)
Behavioral: Therapy — Non-directive therapy performed by a team of two co-therapists

SUMMARY:
This study will examine MDMA-assisted psychotherapy in individuals aged 18 years or older diagnosed with PTSD, with PTSD symptoms not improving after trying at least one treatment. This objective of this study is to determine whether three eight-hour long sessions of MDMA-assisted psychotherapy, scheduled three to five weeks apart, can be safely administered to participants with PTSD, and whether combining a fully therapeutic dose of MDMA with psychotherapy, when compared with a low ("active placebo") dose of MDMA, will reduce PTSD symptoms. Participants will be randomly assigned to receive the full dose of MDMA (125 mg) or assigned to receive a low or "active placebo" dose of MDMA (25 mg) during each of three experimental sessions.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) occurs after experiencing a traumatic event or events. PTSD is a public health problem that causes a great deal of suffering.

This study will examine MDMA-assisted psychotherapy in individuals aged 18 years or older diagnosed with PTSD, with PTSD symptoms not improving after trying at least one treatment. This objective of this study is to determine whether three eight-hour long sessions of MDMA-assisted psychotherapy, scheduled three to five weeks apart, can be safely administered to participants with PTSD, and whether combining a fully therapeutic dose of MDMA with psychotherapy, when compared with a low ("active placebo") dose of MDMA, will reduce PTSD symptoms. Participants will be randomly assigned to receive the full dose of MDMA (125 mg) or assigned to receive a low or "active placebo" dose of MDMA (25 mg) during each of three experimental sessions.

People who receive the low dose of MDMA have the opportunity to take part in a second "open label" study continuation, wherein the participants will undergo three MDMA-assisted sessions, with the participant and the researchers knowing that a full dose of MDMA is being administered. People who receive the full dose of MDMA, and any person who received low-dose MDMA and does not undergo the open-label study continuation will have PTSD symptoms measured six and twelve months after the third session. People who take part in the open label study continuation have their PTSD symptoms assessed six and 12 months after the third Phase II MDMA-assisted session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with posttraumatic stress disorder (PTSD).
* PTSD still remains after one or more prior treatment, with treatment including psychotherapy (talk therapy) or drug therapy
* May meet criteria for a mood disorder
* Must be at least 18 years old
* Must be able to stop taking psychiatric medication during the course of the study, from the start of the study to the follow-up two months after experimental session 3.
* Must agree to follow all rules and instructions relating to the experimental session, including restrictions on food and substance (alcohol and drug) consumption.
* Must be willing to stay overnight at the researcher's office after each experimental session until the non-drug session occurring the next morning.
* Must be willing to be contacted by one of the researchers on a daily basis for a week after each experimental session.
* Female participants of childbearing potential must have a negative pregnancy test and must agree to use an effective form of birth control.
* Participants must have sufficient proficiency in speaking the German language to participate in MDMA-assisted psychotherapy. Participants must be able to read documents in German.

Exclusion Criteria:

* Cannot have history of or current primary psychotic disorder or bipolar affective disorder-1.
* Dissociative identity disorder, or an eating disorder with active purging or borderline personality disorder.
* Evidence or history of significant hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder. (People with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded).
* Uncontrolled hypertension, peripheral vascular disease, hepatic disease (with or without abnormal liver enzymes), or history of hyponatremia or hyperthermia.
* Being pregnant or lactating (nursing), or not practicing an effective method of birth control.
* Weight of less than 50 or more than 105 kg.
* Patients reporting prior use of "Ecstasy" more than 5 times or at any time within the previous 6 months.
* People who would present a serious suicide risk or who are likely to require hospitalization during the course of the study.
* People who need ongoing concomitant therapy with a psychotropic drug.
* Meeting DSM-IV criteria for substance abuse or dependence for any substance save caffeine or nicotine in the past 60 days.
* People who cannot give adequate consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-09-13 (Actual); Primary Completion 2009-09-02 (Actual); Study Completion 2011-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Oehen, MD, Principal Investigator — private practice, Biberist, Switzerland
Locations (1):
- Offices of Peter Oehen MD, Biberist, Canton of Solothurn, Switzerland

REFERENCES:
- [Result] Oehen P, Traber R, Widmer V, Schnyder U. A randomized, controlled pilot study of MDMA (+/- 3,4-Methylenedioxymethamphetamine)-assisted psychotherapy for treatment of resistant, chronic Post-Traumatic Stress Disorder (PTSD). J Psychopharmacol. 2013 Jan;27(1):40-52. doi: 10.1177/0269881112464827. Epub 2012 Oct 31. PMID 23118021
- [Derived] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Derived] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Derived] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by calling for referrals from psychiatric hospitals, trauma counseling centers, psychiatrists and psychotherapists in the German-speaking part of Switzerland.
Pre-assignment Details: Only active control participants from Stage 1 entered into open-label Stage 2 and only participants who received full dose in Stage1 or Stage 2 and did not respond with significant improvement were offered the opportunity to partake in open-label Stage 3.
Groups:
- Full Dose MDMA-assisted Therapy (125 mg Stage 1): Three 8-hour sessions of MDMA-assisted therapy with 125 mg of MDMA, followed by a supplemental dose of 62.5 mg MDMA
  3,4-methylenedioxymethamphetamine (125 mg): Participants will receive an initial dose of 125 mg MDMA orally and, if investigator and participant deem appropriate, 2.5 hours later they will receive 62.5 mg MDMA orally.
  Therapy: Non-directive therapy performed by a team of two co-therapists
- Active Placebo MDMA-assisted Therapy (25 mg Stage 1): Three 8-hour sessions of MDMA-assisted therapy with 25 mg of MDMA, followed by a supplemental dose of 12.5 mg MDMA
  3,4-methyelendioxymethamphetamine (25 mg): Participants will receive a 25 mg MDMA orally, and if investigator and participant agree, 2.5 hours later they will receive 12.5 mg MDMA orally.
  Therapy: Non-directive therapy performed by a team of two co-therapists
- Full Dose MDMA-assisted Therapy (125 mg Stage 2): Three 8-hour sessions of MDMA-assisted therapy with 125 mg of MDMA, followed by a supplemental dose of 62.5 mg MDMA
  3,4-methylenedioxymethamphetamine (125 mg): Participants will receive an initial dose of 125 mg MDMA orally and, if investigator and participant deem appropriate, 2.5 hours later they will receive 62.5 mg MDMA orally.
- Full or Larger Dose MDMA-assisted Therapy (125 or 150 mg Stage 3): Two 8-hour sessions of MDMA-assisted therapy with 125 mg of MDMA, followed by a supplemental dose of 62.5 mg MDMA, or a 20% larger dose of 150 mg MDMA, followed by a supplemental dose of 75 mg administered 2.5 hours later.
  3,4-methylenedioxymethamphetamine (125 or 150 mg): Participants will receive an initial dose of 125 mg MDMA orally and, if investigator and participant deem appropriate, 2.5 hours later they will receive 62.5 mg MDMA orally or Participants will receive an initial dose of 150 mg MDMA orally and, if investigator and participant deem appropriate, 2.5 hours later they will receive 75 mg MDMA orally.
Period: Overall Study
Arm/Group | Full Dose MDMA-assisted Therapy (125 mg Stage 1) | Active Placebo MDMA-assisted Therapy (25 mg Stage 1) | Full Dose MDMA-assisted Therapy (125 mg Stage 2) | Full or Larger Dose MDMA-assisted Therapy (125 or 150 mg Stage 3)
Started | 9 | 5 | 0 | 0
Completed Stage 2 | 0 | 0 | 4 | 0
Completed Stage 3 | 0 | 0 | 0 | 3
Completed (Completed Stage 1) | 8 | 5 | 0 | 0
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Dose MDMA-assisted Therapy (125 mg) | Active Placebo MDMA-assisted Therapy (25 mg) | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (12.8) | 40.0 (6.2) | 41.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Country of origin [Count of Participants; unit: Participants]
  Switzerland | 7 | 4 | 11
  France | 1 | 0 | 1
Work status [Count of Participants; unit: Participants]
  On disability | 4 | 1 | 5
  Fit for limited employment | 2 | 1 | 3
  Working full-time | 1 | 2 | 3
  Retired | 1 | 0 | 1
Duration of PTSD [Mean (Standard Deviation); unit: years] | 16.4 (10.9) | 22.3 (12.1) | 18.3 (12.0)
Duration of prior therapy [Mean (Standard Deviation); unit: months] | 39.9 (73.3) | 123 (60.6) | 85.8 (71.4)
On medication for PTSD at enrollment [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 6
  No | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Primary Endpoint in Clinician Administered PTSD Scale for DSM-IV (CAPS-IV)
Description: The CAPS-IV is a structured clinical interview designed to assess the symptoms and severity of PTSD. The CAPS-IV provides a means to evaluate the frequency and intensity dimensions of each symptom, the impact of symptoms on the patient's social and occupational functioning, the overall severity of the symptom complex, global improvement since baseline, and the validity of the ratings obtained. Total severity scores range from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Less than 4 weeks before first experimental session (Baseline) to 3 weeks post 3rd experimental session (Primary Endpoint)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Dose MDMA-assisted Therapy (125 mg) | Active Placebo MDMA-assisted Therapy (25 mg)
Number analyzed (Participants) | 8 | 4
score on a scale | -15.6 (18.1) | 3.3 (15.3)

2. Secondary Outcome: Change From Baseline to Primary Endpoint in Posttraumatic Stress Diagnostic Scale (PDS)
Description: The Posstraumatic Stress Diagnostic Scale (PSD) is a 49-item self-report instrument to aid in the diagnosis of PTSD. Questions are asked about symptoms experienced and participants respond on a scale from 0 ("not at all or only one time") to 3 ("5 or more times a week/almost always"). Items are summed to create a total score that ranges from 0 to 51, with higher scores indicating more PTSD symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Dose MDMA-assisted Therapy (125 mg) | Active Placebo MDMA-assisted Therapy (25 mg)
Number analyzed (Participants) | 8 | 4
score on a scale | -8.6 (13.0) | 7.3 (6.2)

ADVERSE EVENTS:
Time Frame: From baseline to end of Stage 3 (approximately 1 year)
Arm/Group | Full Dose MDMA-assisted Therapy (125 mg Stage 1) | Active Placebo MDMA-assisted Therapy (25 mg Stage 1) | Full Dose MDMA-assisted Therapy (125 mg Stage 2) | Full or Larger Dose MDMA-assisted Therapy (125 or 150 mg Stage 3)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 8/9 | 3/5 | 2/4 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Dose MDMA-assisted Therapy (125 mg Stage 1) (N=9) | Active Placebo MDMA-assisted Therapy (25 mg Stage 1) (N=5) | Full Dose MDMA-assisted Therapy (125 mg Stage 2) (N=4) | Full or Larger Dose MDMA-assisted Therapy (125 or 150 mg Stage 3) (N=3)
Metasteses to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Suicidal behavior (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Full Dose MDMA-assisted Therapy (125 mg Stage 1) (N=9) | Active Placebo MDMA-assisted Therapy (25 mg Stage 1) (N=5) | Full Dose MDMA-assisted Therapy (125 mg Stage 2) (N=4) | Full or Larger Dose MDMA-assisted Therapy (125 or 150 mg Stage 3) (N=3)
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 2 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Psychiatric disorders) | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia chlamydial (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Somnolence (Psychiatric disorders) | 1 | 0 | 0 | 0
Tension (Psychiatric disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Nervous system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0
Iron deficiency Anemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Angina tonsillitus (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2010-01-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT00353938/Prot_001.pdf
  • Statistical Analysis Plan (2011-05-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT00353938/SAP_002.pdf
  • Informed Consent Form (2007-12-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT00353938/ICF_000.pdf